CLINICAL TRIAL: NCT06424392
Title: Respiratory and Psychological Impact of Elective Surgery of Congenital Lung Malformations
Acronym: MALFPULM2
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-A00576-41
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Congenital Lung Malformations
Keywords: Congenital lung malformations; Psychological impact

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 6-9 years children with their parent(s)with fetal diagnoses of CLM: 6-9 years children with their parent(s) with fetal diagnoses of CLM and included in MALFPULM who have had at least one follow-up visit between 0 and 2 years of age.
  Interventions: Other: General Health Questionnaire (GHQ-12); Other: State-Trait Anxiety Inventory (STAI-Y); Other: Revised Children's Manifest Anxiety Scale (RCMAS); Other: World Health Organization Quality of Life (WHOQOL-BREF); Other: Parental Educational Competence Self-Evaluation Questionnaire "Questionnaire d'Auto-Évaluation de la Compétence Éducative Parentale (QAECEP)"; Other: Parental interview

INTERVENTIONS:
Other: General Health Questionnaire (GHQ-12) — Anxiety and depression self-reported scales for both parents
Other: State-Trait Anxiety Inventory (STAI-Y) — Anxiety and depression self-reported scales for both parents
Other: Revised Children's Manifest Anxiety Scale (RCMAS) — Anxiety and depression self-reported scales for children
Other: World Health Organization Quality of Life (WHOQOL-BREF) — Quality of life self-reported scales for parents
Other: Parental Educational Competence Self-Evaluation Questionnaire "Questionnaire d'Auto-Évaluation de la Compétence Éducative Parentale (QAECEP)" — Parental Educational Competence Self-Evaluation self-reported Questionnaire for parents
Other: Parental interview — The interview will only last about ten minutes and will take place during the first call, if the parents have agreed and are sufficiently available to answer. If the parents are not available, an appointment can be made at a later date

SUMMARY:
The absence of surgery of Congenital lung malformations (CLMs), if it avoids a stressfull event, is accompanied by a "medicalization" of the child, which will be regularly followed up in a specialized medical and surgical environment. The persistent risk of complication, albeit low, is likely to induce over-protective parental behaviours, and to be associated with a sustained family anxiety reaction. The main objective is to test the hypothesis that the absence of surgery has a significant impact on parental anxiety, measurable at 6- 9 years of age.

DETAILED DESCRIPTION:
The knowledge of CLMs has been revolutionized by prenatal imaging and the identification of large numbers of CLMs that remain asymptomatic. France is a leader in this field, having set up the only prospective multicentre cohort currently available internationally, with follow-up starting in the prenatal period (MALFPULM). This cohort has already enabled a better description of the prenatal history and the development of an algorithm predictive of the risk of neonatal respiratory distress. The children were followed up to the age of 2 years, and 66% of them were operated on between 0 and 2 years of age. This cohort is a unique opportunity to measure the mid-term impact of this surgical decision, in terms of both medical complications and psychological consequences.

In particular, the size of the cohort makes it possible to answer with a sufficient level of evidence to the following controversies:

* What is the risk of CLM infection in the absence of surgical removal, and is this risk dependent on the CLM phenotype?
* What is the functional respiratory impact of surgical techniques (thoracoscopy or thoracotomy), depending on the age of the surgery?
* What is the prevalence of musculoskeletal complications according to surgical techniques (thoracoscopy or thoracotomy)?
* What is the burden of the medical or surgical follow-up depending on the chosen therapeutic option?
* What is the psychological impact of the surgical decision on the parents and the child? Considering the psychological impact is a major issue for this malformative condition which mainly concerns asymptomatic children, and is of great originality because it has never been evaluated. The most recent literature clearly calls for integrating issues of family well-being and parental mental health into the follow-up of children with chronic disease and/or congenital anomalies. For this reason, the investigators chose maternal anxiety as the main criterion of this study. Specifically for CLM, demonstrating the impact of the investigator's decisions on the psychological state of the parents will be a strong encouragement to integrate this dimension in care, for a better detection of these anxious and/or depressive parental reactions, and a better personalization of the transmission of decisions.

ELIGIBILITY:
Inclusion Criteria:

* Child of the MALFPULM cohort, with their parents
* At least one follow-up visit between 0 and 2 years of age (n= 414 eligible children)
* Non-opposition of the family

Exclusion Criteria:

* Child with CLM, but not included in MALFPULM
* Parents who participated in MALPULM, but with prenatal fetal death, or neonatal death.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The families of all children included in MALFPULM who have had at least one follow-up visit between 0 and 2 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 434 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
maternal anxiety level | 1 year
  The level of maternal anxiety is measured using the GHQ-12 anxiety scale. The GHQ ( General Health Questionnaire) consists of 12 items, each assessing the severity of a mental problem over the past few weeks. Each reponse is scored from 0 to 3, with a total score ranging from 0 to 36. Higher scores indicate poorer health.

SECONDARY OUTCOMES:
Impact of the surgical decision on respiratory morbidity - lower respiratory tract infections | 1 year
  Number of lower respiratory tract infections, either documented (radiological opacity) or not, in the last 12 months and from birth to the date of evaluation
Impact of the surgical decision on respiratory morbidity - hospitalizations | 1 year
  Number of hospitalizations for respiratory reasons in the last 12 months and from birth to the date of evaluation
Impact of the surgical decision on respiratory morbidity - severe wheezing respiratory exacerbations | 1 year
  Number of severe wheezing respiratory exacerbations in the last 12 months, defined as requiring oral corticosteroids, emergency visit and/or hospitalization
Impact of the surgical decision on respiratory morbidity - treatment | 1 year
  Current regular treatment for respiratory purposes, defined as daily treatment for at least 3 consecutive months in the last 12 months
Impact of the surgical decision on respiratory morbidity - lung function tests | 1 year
  Following parameters will be collected: date of performance, weight and height at date of performance, total lung capacity (TLC), forced vital capacity (FVC), forced expiratory volume in one second (FEV1), Forced expiratory flow at 25-75% (FEF25-75%), transfer factor of the lung for carbon monoxide (TLCO). FVC, FEV1, and FEF25-75%. These measurements will allow to identify following functional profiles:
  * lung function restriction, defined by TLC lower than -1.645 Z score
  * airway obstruction, defined by FEV1/FVC lower than -1.645 Z score, and its reversibility, defined by an improvement of at least 12% of the FV1 after inhalation of salbutamol.
  * impaired diffusion capacity, defined by DLCO lower than -1.645 Z score.
Impact of the surgical decision on respiratory morbidity - thoracic deformities | 1 year
  The parents's declare rate of thoracic deformities
Impact of the surgical decision on respiratory morbidity - burden of the medical or surgical follow-up | 1 year
  The burden of the medical or surgical follow-up will be evaluated by the number of specialist consultations and the number of CT or MRI scans
Anxiety and depression - GHQ-12 | 1 year
  The 12-item GHQ (General Health Questionnaire) was designed to be a self-administered screening test aimed at detecting minor psychiatric disorders and had been and validated in different languages, including French. It allows to estimate the prevalence of psychological distress in a given population (34). The GHQ-12 consists of 12 items, each one assessing the severity of a mental problem over the past few weeks, with four response options, and using six positively phrased and six negatively phrased. It takes less than 5 minutes to complete. It is scored from 0 to 3 for each response with a total possible score on the ranging from 0 to 36. High scores indicate worse health.
Anxiety and depression - STAI-Y | 1 year
  The State-Trait Anxiety Inventory (STAI-Y) is a 20-item self-measure of state anxiety level in parents, complementary of GHQ-28. It reflects the current subjective feeling of tension, apprehension, nervousness, and worry and is widely used both in practice and in clinical research.
Anxiety and depression - RCMAS | 1 year
  The RCMAS is a 37-item, self-report instrument designed to assess the level and nature of anxiety. A Total Anxiety score is computed based on 28 items, which are divided into three anxiety subscales: physiological anxiety (10 items about somatic manifestations of anxiety such as sleep difficulties, nausea and fatigue), worry/oversensitivity (11 items measuring obsessive concerns about a variety of things, most of which are typically vague and ill-defined, as well as fears about being hurt or emotionally isolated), and social concerns/concentration (7 items measuring distracting thoughts and fears that have a social or interpersonal nature). The remaining nine items on the RCMAS constitute the Lie subscale. A high score indicates a high level of anxiety or lie on that subscale.
Quality of life - WHOQOL-BREF | 1 year
  The WHOQOL-BREF is an abbreviated form of the WHOQOL-100 with only 26 items. It is an instrument for recording subjective quality of life. This is defined as an individual perception of one's own life situation in the context of culture and value system as well as personal goals, expectations, evaluation criteria and interests. It is a self-questionnaire that includes the four domains "physical health", "psychological well-being", "social relationships" and "environment". The items are answered using a five-level scale. The scales have a very high internal consistency. It is validated in several languages, including French.
Parenting Sense of Competence questionnaire | 1 year
  This questionnaire evaluates the parent's sense of competence in his or her role as an educator and has two components: the "skill/knowledge" factor, which evaluates the respondents' perception of the skills and knowledge they have acquired in order to be adequate parents (8 items); the "value/ease" factor, which evaluates the value that the respondent places on the role of parent, as well as his or her ease in this role (9 items).
Over-protective parental behaviours | 1 year
  The over-protective parental behaviours is defined by the age of attendance in first community (5 or more children), the care arrangements between 0 and 2 years, the after-school activities in the previous year and the travel outside France in the last two years

CONTACTS AND LOCATIONS:
Overall Officials: Christophe DELACOURT, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No